CLINICAL TRIAL: NCT02377674
Title: To Assess the Initial Safety and Performance of COR-VG-001 Conduit in Pediatric Patients Undergoing Extracardiac Total Cavopulmonary Connection (EC-TCPC)
Brief Title: Safety and Performance of the COR-VG-001 Conduit in Pediatric Patients for Extracardiac Total Cavopulmonary Connection
Acronym: EC-TCPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Collaborators: Technomics Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-05
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Vascular Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vascular Graft, Model COR-VG-001 (Experimental): A surgically implanted vascular graft for pediatric patients undergoing extracardiac total cavopulmonary connection.
  Interventions: Device: Vascular Graft, Model COR-VG-001

INTERVENTIONS:
Device: Vascular Graft, Model COR-VG-001 — The intended use of the Xeltis Vascular Graft, Model COR-VG-001 is to create an extracardiac total cavopulmonary connection (EC-TCPC) connection to divert the venous blood from the inferior vena cava to the pulmonary arteries without passing through the morphologic right ventricle reducing the volume load on the functional single ventricle and thereby improving hemodynamics by minimizing the deleterious effects of ventricular hypertrophy.

SUMMARY:
The extracardiac Fontan surgery/procedure involves diverting the venous blood from the inferior vena cava to the pulmonary arteries without passing through the morphologic right ventricle. In the extracardiac conduit type of Fontan, one end of a synthetic tube graft is connected to the inferior vena cava and the other end to the pulmonary artery confluence.

Xeltis developed a biodegradable prosthesis, the Xeltis Vascular Graft Model COR-VG-001, to be used as an extracardiac conduit between right atrium and the pulmonary arteries. The prosthesis is immediately mechanically functional, while its physiochemical characteristics should enable cell infiltration and tissue formation.

The Xeltis Vascular Graft Model COR-VG-OO is specifically designed to enhance the Fontan surgery outcome by reducing synthetic material related complications and improving hemodynamic characteristics.

DETAILED DESCRIPTION:
Although significant progress has been made in recent years in the field of congenital heart disease treatment, a substantial unmet clinical need remains for implantable materials/devices such as vascular grafts and heart valves with improved long-term performance and reduced device-related complications.

To address these limitations new generation of biodegradable polymers using recent advances in supramolecular chemistry have been developed to create highly porous vascular grafts allowing efficient cell infiltration following by gradual replacement of the polymer material with the patient's own native-like vascular tissue resulting in full functional restoration. In addition to the ability of reducing postoperative graft-related complications such types of implants have a potential to grow to adapt to the overall body growth and therefore may represent a completely new modality for the treatment of congenital heart disease. In contrast to today's situation with synthetic non-absorbable vascular grafts considered as a "standard of care", where the pediatric patients have to be re-operated several times to adjust the prosthesis size to the somatic growth of the child associated with substantial morbidity and mortality and requiring prolonged anticoagulation treatment, a biodegradable polymer implant could represent a "one-time solution".

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring EC-TCPC
2. Male or Female
3. Aged ≥ 2 years

Exclusion Criteria:

1. Pulmonary artery pressure (PAP) > 15 mm Hg as excluded by angiography/cardiac catheterization
2. Pulmonary vascular resistance (PVR) >3 Wood units as excluded by angiography/cardiac catheterization
3. Moderate or severe atrioventricular (AV) valve regurgitation requiring correction, as determined by echocardiography and/or angiography
4. Moderate or severe outflow valve regurgitation requiring correction as determined by echocardiography and/or angiography
5. Outflow tract (aortic arch and isthmus) obstruction as excluded by:

   * a residual outflow gradient of ≥ 20mm Hg or
   * requirement of corrective surgery
   * as determined by echocardiography and/ or angiography
6. All arrhythmias as determined by ECG and/or at the investigator's discretion
7. Renal dysfunction as excluded by serum creatinine > ULN and/or urea >ULN and/or at the investigator's discretion
8. Hepatic dysfunction as excluded by ALT >ULN, AST > ULN, GGT > ULN and/or at the investigator's discretion
9. Coagulation disorders as defined by INR outside its normal value, PTT >ULN and Fibrinogen <LLN and/or at the investigator's discretion
10. Transcutaneous O2 saturation < 65% and/or at the investigator's discretion
11. Immunodeficiency
12. Trisomia 21
13. Asplenia as determined by abdominal ultrasound
14. Heterotaxia as determined by abdominal ultrasound
15. HIV-infection
16. Syphilis (Treponema pallidum)
17. Hepatitis-B and/or -C virus infection
18. Unwillingness of Parental/legal guardian to give consent
19. Contraindications on ethical grounds
20. Treatment with other investigational products
21. Known or suspected non-compliance, drug or alcohol abuse of the parents/legal guardian
22. Inability of the parents/legal guardian to follow the procedures of the study, e.g. due to language problems
23. Participation of the patient in another study within 30 days preceding and during the present study
24. Previous enrollment of the patient into the current study
25. Enrollment of the investigator's family members, employees and other dependent persons

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Bockeria, Professor, Principal Investigator — Bakoulev Center of Cardiovascular Surgery
Locations (1):
- Bakoulev Center of Cardiovascular Surgery, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vascular Graft, Model COR-VG-001
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vascular Graft, Model COR-VG-001
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.2 [4 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Graft Related Post-operative Complications That Require a Repeat Surgery or a Non Surgical Treatment Within 12-month Post Implantation.
Description: Evaluation of the safety of the COR-VG-001 as defined by numbers of patients having graft related post-operative complications requiring surgery, intervention or leading to death within 12-month post implantation
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vascular Graft, Model COR-VG-001
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: The Number of Grafts That Have a Reduced Function Post Operatively.
Description: Evaluation of the performance of the COR-VG-01 by analyzing, with the help of echocardiography, the incidence of loss of functionality requiring intervention within 12 months post implantation.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vascular Graft, Model COR-VG-001
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Arm/Group | Vascular Graft, Model COR-VG-001
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascular Graft, Model COR-VG-001 (N=5)
Left Lower Lobe Pneumonia (Infections and infestations) | 1 (1)
Pleural Effusion Caused by Cardiac Failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cardiac Failure, poly seriositis NYHA III (Cardiac disorders) | 1 (1)
Stenosis of Conduit (Product Issues) | 1 (1)
Decreased LVEF (Cardiac disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascular Graft, Model COR-VG-001 (N=5)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1)
Bundle Branch Block Onset (Cardiac disorders) | 1 (1)
Decreased Ejection Fraction (Cardiac disorders) | 1 (1)
Low Stroke Volume in the IVC and Conduit (Cardiac disorders) | 1 (1)
Cold (Infections and infestations) | 2 (2)
Mild Stenosis In Conduit (Cardiac disorders) | 1 (1)
Reduced Maximum Systolic Velocity (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Researchers engaged in Project can present research results provided the Sponsor has been furnished copies at least one month in advance of the submission. Sponsor shall have thirty (30) days, after receipt of said copies, to object because there is confidential subject matter or proprietary information of Sponsor which needs protection. In the event that Sponsor makes such objection, said Researcher(s) shall refrain from making such publication or presentation for a maximum of six months